CLINICAL TRIAL: NCT02636998
Title: Nutrition and Cognitive Function in Preadolescents
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 204071
Record Dates: First submitted 2015-06-22; First posted 2015-12-22 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2024-09

CONDITIONS: Healthy Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and salivary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight: BMI <85th percentile
- Obese: BMI > 95th percentile

SUMMARY:
This study is designed to evaluate cognitive function in preadolescents who have different body mass indexes.

DETAILED DESCRIPTION:
The investigators plan to document differences between normal weight and obese preadolescents on psychological and neurocognitive measures of executive function controlling for factors known to influence brain function and behavior not considered in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI: <85th percentile) or obese (BMI: >95th percentile)
* Right hand dominance
* Report eating breakfast at least 4 days/week
* Able to hear at least 20 dB stimulus
* Visual acuity must be at least 20/40
* Arithmetic Computation Task
* Biological mother available to attend the enrollment study visit

Exclusion Criteria:

* Full Scale IQ <80
* Children taking medications or having chronic illnesses/disorders that may independently affect study outcome measures (as determined by the PI)

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preadolescents and their mothers
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Psychological assessments | 9-10 years
  Standardized assessments
Neurocognitive measures | 9-10 years
  Brain Lab Recordings

CONTACTS AND LOCATIONS:
Overall Officials: Linda Larson-Prior, Ph.D, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

DOCUMENTS (1):
  • Informed Consent Form (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT02636998/ICF_001.pdf